CLINICAL TRIAL: NCT03933566
Title: Comparison Between Ultrasound-Guided and Landmark-Based Superficial Cervical Plexus Block：A Retrospective Observational Study
Brief Title: US-Guided Superficial Cervical Plexus Block
Status: Completed | Type: Observational
Sponsor: Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2019CZTCWM2
Record Dates: First submitted 2017-12-29; First posted 2019-05-01 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2019-04

CONDITIONS: Nerve Block
Keywords: Ultrasound-Guided Superficial Cervical Plexus Block; Landmark-Based Superficial Cervical Plexus Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound-Guided: Ultrasound-Guided Superficial Cervical Plexus Block
  Interventions: Procedure: Ultrasound-Guided Superficial Cervical Plexus Block
- Landmark-Based: Landmark-Based Superficial Cervical Plexus Block
  Interventions: Procedure: Landmark-Based Superficial Cervical Plexus Block

INTERVENTIONS:
Procedure: Ultrasound-Guided Superficial Cervical Plexus Block — Ultrasound-Guided Superficial Cervical Plexus Block
  Groups: Ultrasound-Guided
Procedure: Landmark-Based Superficial Cervical Plexus Block — Landmark-Based Superficial Cervical Plexus Block
  Groups: Landmark-Based

SUMMARY:
This retrospective observational study compare ultrasound-guided plane and landmark-based superficial cervical plexus block

DETAILED DESCRIPTION:
Traditionally, the superficial cervical plexus is blocked using a subcutaneous infiltration of local anesthetics along the posterior border of the sternocleidomastoid muscle.Recently, ultrasound has been used to identify intermuscular planes to carry out transversus abdominis plane and obturator nerve blocks.Thus, to validate this new method, the investigators conducted a retrospective observational study comparing ultrasound and the conventional landmark-based technique for superficial cervical plexus.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery of the shoulder and clavicle
* Urgent or planned surgery

Exclusion Criteria:

* Refused to sign informed consent
* Pregnant women
* Allergic to the local anesthetic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Success rate | At 15 mins after nerve block
  Number of Participants wit absence of pain sensation for all 4 branches of the superficial cervical plexus

CONTACTS AND LOCATIONS:
Overall Officials: Ruizhao Lv, M.D, Principal Investigator — Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine
Locations (1):
- Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided